CLINICAL TRIAL: NCT04271475
Title: A Prospective, Randomized, Double-blind, Multicenter, Placebo-controlled, Parallel Group, Adaptive Phase 3 Study With Open-label Extension to Evaluate Efficacy and Safety of Macitentan 75 mg in Inoperable or Persistent/Recurrent Chronic Thromboembolic Pulmonary Hypertension
Brief Title: A Study to Evaluate Efficacy and Safety of Macitentan 75 mg in Inoperable or Persistent/Recurrent Chronic Thromboembolic Pulmonary Hypertension
Acronym: MACiTEPH
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Sponsor decided to stop the study for futility based on a recommendation by the IDMC following a pre-planned interim analysis
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108742; 67896062CTP3001 (Other: Janssen Research & Development, LLC); 2019-004131-24 (EudraCT Number)
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
MeSH Terms: interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Macitentan (Experimental): Participant will receive macitentan at a dose of 10 milligram (mg) once daily (OD) for 4 weeks, followed by a dose of macitentan 37.5 mg for another 4 weeks and continue with the target dose of macitentan 75 mg. Participants who have reached the target dose of 75 mg, completed the Double-blind (DB) period up to Week 28 (either on treatment or in Post-treatment observation period [PTOP]) at minimum, may be eligible for transitioning into the Open label (OL) extension period once all participants have completed the DB part of the study, or earlier if they experienced a Clinical event committee (CEC) confirmed clinical worsening event.
  Interventions: Drug: Macitentan
- Placebo (Experimental): Participants will receive placebo tablets matching the macitentan 10 mg, macitentan 37.5mg and macitentan 75 mg tablets, respectively. Participants who completed the DB period as per protocol either on treatment or in PTOP are eligible for transitioning to the OL extension period and will receive macitentan 75 mg after an 8-week double-dummy uptitration (macitentan 10 mg for 4 weeks, followed by 37.5 mg for another 4 weeks).
  Interventions: Drug: Macitentan; Drug: Placebo

INTERVENTIONS:
Drug: Macitentan — Participants will receive Macitentan film-coated tablets orally od.
  Other Names: ACT-064992,; Opsumit
Drug: Placebo — Participant will receive matching placebo tablets orally od.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the effect of macitentan 75 mg versus placebo on exercise capacity at Week 28 in participants with chronic thromboembolic pulmonary hypertension (CTEPH).

DETAILED DESCRIPTION:
CTEPH is one of the leading causes of severe pulmonary hypertension (PH), classified within World Health Organization (WHO) group 4 PH. It is a rare, progressive pulmonary vascular disease that if left untreated, leads to progressively increasing pulmonary vascular resistance (PVR) and eventually right ventricle failure and death. Histopathologic findings including endothelial cell dysfunction and distal pulmonary arterial remodeling are shared between PAH and CTEPH, and PH-specific therapies (that is, riociguat) have shown efficacy in inoperable and persistent/recurrent CTEPH. The endothelin receptor antagonist macitentan offers a different mode of action and addresses an important unmet medical need for an alternative treatment option in this indication. This study will assess the effect of macitentan 75 mg on exercise capacity in CTEPH. The total duration of the study is approximately 6 years. The study comprises of a screening period (at least 14 days and up to 60 days), a double-blind (DB) treatment period (28 weeks [minimum duration] up to 3.5 years), an open-label (OL) extension period (starts at end-of-DB-treatment [EODBT] and will end for all participants 104 weeks after the last participant has completed DB Week 28). The DB period consists of an 8-week up-titration phase and a maintenance phase. The maintenance phase is divided into a 28-week fixed duration part, at the end of which primary endpoint is assessed, and a variable duration part. The duration of the DB period for an individual participant depends on the timepoint of entry into the study and whether a CEC-confirmed clinical worsening event occurred. Participants who discontinue DB study intervention during the 28-week fixed duration part will be followed until Week 28 in a post-treatment observation period (PTOP).

ELIGIBILITY:
Inclusion Criteria:

* Chronic thromboembolic pulmonary hypertension (CTEPH) (World Health Organization [WHO] Group 4) fulfilling one of the following criteria: a) inoperable due to the localization of the obstruction being surgically inaccessible (that is, distal disease), b) persistent/recurrent CTEPH after balloon pulmonary angioplasty (BPA), and deemed inoperable due to the localization of the obstruction being surgically inaccessible (that is, distal disease), c) persistent/recurrent CTEPH after rescue pulmonary endarterectomy (PEA)
* 6-minute walk distance (6MWD) greater than or equal to (>=) 100 meter (m) and less than or equal to (<=) 450 meters (m), documented by an eligibility and a baseline 6-minute walk test (6MWT). The baseline 6MWD must not differ by more than 15 percent (%) from the eligibility test
* World Health Organization functional class (WHO FC) >= II
* Participants are to receive riociguat as per local standard of care, unless it is contraindicated or unavailable

Exclusion Criteria:

* Acute pulmonary embolism within 3 months prior to or during Screening
* Planned balloon pulmonary angioplasty (BPA) during the fixed duration part of the double-blind period
* Significant obstructive and restrictive lung disease
* Acute or chronic conditions (other than dyspnea) that limit the ability to comply with study requirements, in particular with 6MWT (for example, intermittent claudication).
* Symptomatic coronary artery disease requiring an intervention within 3 months prior to or during Screening or anticipated during the fixed duration part of the study
* Decompensated cardiac failure if not under close supervision
* Known and documented life-threatening cardiac arrhythmias
* Acute myocardial infarction within 6 months prior to, or during Screening
* Cerebrovascular events (including transient ischemic attack) within 3 months prior to, or during Screening
* Known or suspicion of pulmonary veno-occlusive disease (PVOD)
* Administration of ERAs, intravenous prostacyclins / prostacyclin analogs, or investigational treatment within 90 days prior to Randomization
* Change in dose or initiation of Phosphodiesterase type-5 (PDE-5) inhibitors, oral, inhaled or subcutaneous (SC) prostacyclins / prostacyclin analogues, prostacyclin receptor agonists or riociguat, a) within 90 days prior to Randomization, or b) anticipated during the fixed duration part of the double-blind [DB] period
* Hypotension, that is, systolic blood pressure (SBP) less than (<) 90 millimeters of mercury (mmHg) or diastolic blood pressure (DBP) <50 mmHg at Screening.
* Severe renal dysfunction with an estimated Glomerular Filtration Rate <30 milliliters per minute per 1.73 meter square (mL/min/1.73 m^2) using the Chronic Kidney Disease Epidemiology Collaboration formula at Screening
* Known moderate to severe hepatic impairment, defined as Child-Pugh Class B or C, based on records that confirm documented medical history
* Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) greater than or equal to (>=) 1.5*upper limit of normal (ULN) at Screening
* Hemoglobin <100 g/L (<10 gram per deciliter [g/dL]) at Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trial, Study Director — Actelion
Locations (168):
- United States (24):
  - University of California San Diego Medical Center, La Jolla, California
  - Keck School of Medicine of USC, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale University School Of Medicine, New Haven, Connecticut
  - University of Florida Health Jacksonville, Gainesville, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - University of Nebraska Medical Center, Omaha, Nebraska
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Syracuse VA Medical Center, Syracuse, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Legacy Hospital, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Scott White - Plano, Plano, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Cardiovascular Center, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Argentina (3):
  - Nexo Salud Investigacion Clinica, Buenos Aires
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Sanatorio Guemes, C.a.b.a.
- Australia (2):
  - Queensland Lung Transplant Service, Chermside
  - St Vincent's hospital, Darlinghurst
- Austria (3):
  - LKH-Univ. Klinikum Graz, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Medizinische Universitaet Wien, Vienna
- Bulgaria (2):
  - Military Medical Academy, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
- Canada (3):
  - University Of Calgary - Peter Lougheed Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - University Health Network - Toronto General Hospital, Toronto, Ontario
- China (15):
  - Beijing Chaoyang Hospital, Beijing
  - Beijing Anzhen Hospital, Beijing
  - China Japan Friendship Hospital, Beijing
  - Beijing Shijitan Hospital, Beijing
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - Zhongda Hospital Southeast University, Nanjing
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao
  - Huashan Hospital of Fudan University, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - The General Hospital of Northern Theater Command, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- Colombia (4):
  - Fundacion Neumologica Colombiana, Bogotá
  - Fundación Abood Shaio, Bogotá
  - Clínica Imbanaco S.A.S., Cali
  - Centro Cardiovascular Colombiano Clínica Santa María, Medellín
- General University Hospital II.department of Internal Medicine-cardiology and angiology, Prague, Czechia
- Århus Universitetshospital, Skejby, Hjertemedicinsk Afdeling B, Aarhus N, Denmark
- France (8):
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - CHU de Grenoble Hopital Albert Michallon, Grenoble
  - Hopital Bicetre Aphp Hopitaux Universitaires Paris Sud, Le Kremlin-Bicêtre
  - Hôpital Cardiologique - Chru Lille, Lille
  - CHU de Montpellier - Arnaud de Villeneuve, Montpellier
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Larrey CHU de Toulouse, Toulouse
  - CHU de Nancy - Hopital de Brabois, Vandœuvre-lès-Nancy
- Germany (9):
  - Universitatsklinikum Bonn, Bonn
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Universitaetsklinikum Giessen, Giessen
  - Universitaetsklinikum Hamburg Eppendorf, Hamburg
  - Medizinische Hochschule Hannover Zentrum Innere Medizin Klinik für Pneumologie, Hanover
  - Thoraxklinik Heidelberg, Heidelberg
  - Universitaetsklinikum des Saarlandes, Homburg
  - Universitatsklinikum Jena, Jena
  - Krankenhaus Neuwittelsbach, München
- Hungary (2):
  - Gottsegen Gyorgy Orszagos Kardiovaszkularis Intezet Felnott kardiologiai osztaly, Budapest
  - Szegedi Tudományegyetem, Általános Orvostudományi Kar, Családorvosi Intézet és rendelő, Szeged
- Israel (2):
  - Tel Aviv Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (5):
  - Ospedale SS. Annunziata, Chieti
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio CNR, Pisa
  - Policlinico Gemelli Universita Cattolica, Roma
  - A.O.U. Città della Salute e della Scienza, Torino
- Japan (16):
  - The University of Tokyo Hospital, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Kure Kyosai Hospital, Hiroshima
  - St Marianna University Hospital, Kanagawa
  - Kobe University Hospital, Kobe
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Toho University Medical Center, Ohashi Hospital, Meguro-ku
  - Kyorin University Hospital, Mitaka
  - Nagoya University Hospital, Nagoya
  - National Hospital Organization Okayama Medical Center, Okayama
  - Hokkaido University Hospital, Sapporo
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Juntendo University Hospital, Tokyo
  - University of Tsukuba Hospital, Tsukuba
- Lithuania (2):
  - Lietuvos sveikatos mokslų universiteto ligoninė Kauno klinik, Kaunas
  - Vilnius University Hospital Santariskiu Klinikos, Vilnius
- Mexico (5):
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, Mexico City
  - Operadora de Hospitales Angeles SA de CV Hospital Angeles Lomas, México
  - Unidad de Investigacion Clinica en Medicina S.C. (UDICEM), Monterrey
  - Centro de Investigacion Clinica Chapultepec, Morelia
  - CRI Centro Regiomontano de Investigacion SC, Nuevo León
- Poland (3):
  - Krakowski Szpital Specjalistyczny im Jana Pawla II, Krakow
  - Wojewodzki Szpital Specjalistyczny im Stefana Kardynala Wyszynskiego PZOZ, Lublin
  - Europejskie Centrum Zdrowia Otwock Sp z o o, Otwock
- Uls Almada Seixal - Hosp. Garcia de Orta, Almada, Portugal
- Romania (2):
  - Institutul de urgenta pentru Boli Cardiovasculare Prof. Dr. C.C. Iliescu, Bucharest
  - Spitalul Clinic Judetean de Urgenta, Tg. Mures
- Russia (5):
  - State Autonomous HealthCare Institution 'Interregional Clinical Diagnostic Center', Kazan'
  - Moscow City Clinical Hospital No.51, Moscow
  - National Medical Research Center of Cardiology of MoH of Russian Federation, Moscow
  - National medical Research Center n.a. V.A.Almazov of MoH of Russian Federation, Saint Petersburg
  - Volgograd Regional Clinical Cardiology Center, Volgograd
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - King Fahad Medical City, Riyadh
- Serbia (2):
  - University Clinical Center of Serbia, Belgrade
  - Institute for Pulmonary Disease of Vojvodina, Kamenitz
- Singapore (2):
  - National University Heart Centre, Singapore, Singapore
  - National Heart Centre (NHC) Singapore, Singapore
- Narodny ustav srdcovych a cievnych chorob, Bratislava, Slovakia
- South Korea (5):
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Marys Hospital, Seoul
- Spain (6):
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp Virgen de La Victoria, Málaga
  - Hosp. Costa Del Sol, Málaga
  - Hosp. Gral. Univ. de Toledo, Toledo
- Taiwan (4):
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang-Gung Memorial Hospital, LinKou Branch, Taoyuan District
- Thailand (3):
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Thammasat Hospital, Pathum Thani
- Turkey (Türkiye) (13):
  - Adana City Hospital, Adana
  - Cukurova University Medical Faculty, Adana
  - Hacettepe University Medical Faculty, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Pamukkale University Medical Faculty, Denizli
  - Eskisehir Osmangazi University Medical Faculty Hospital, Eskişehir
  - Istanbul University - Cerrahpasa Cardiology Institution, Istanbul
  - Siyami Ersek Training and Research Hospital, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir
  - Kartal Kosuyolu Yuksek Ihtisas Egitim Ve Arastirma Hastanesi, Kartal Istanbul
  - Mersin University Medical Faculty, Mersin
- Ukraine (6):
  - CNE 'Cherkasy Regional Cardiological Center of Cherkasy Regional Council', Cherkasy
  - CE 'Dnipropetrovsk Regional Clinical Center of Cardiology and Cardiosurgery', Dnipro
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - State Institute Of Phthisiology And Pulmonology N.A. F.G. Yanovskiy Of Ams Ukraine, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council 'Lviv Regional Clinical Hospital', Lviv
  - Municipal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Ternopil
- United Kingdom (6):
  - Papworth Hospital NHS Trust, Cambridge
  - National Waiting Times Centre Board Golden Jubilee National Hospital, Glasgow
  - Royal Free Hospital, London
  - Hammersmith Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study comprised of screening, double-blind (DB), open-label (OL) and safety follow-up (FU) periods. The DB period started with an 8-week up-titration phase and lasted until all participants either completed the Week 28 visit or prematurely discontinued the study.
Groups:
- Double Blind (DB) Period: Macitentan: During the 8-week up-titration phase, participants received macitentan doses orally once daily (QD): 10 mg tablet for 4 weeks followed by 37.5 mg tablet for another 4 weeks prior to reaching the target maintenance phase dose of macitentan 75 mg QD. Participants were to remain on double-blind maintenance treatment until the last participant randomized completed the Week 28 visit. Participants who prematurely discontinued DB study treatment prior to Week 28 but did not withdraw consent were asked to enter post-treatment observation period (PTOP) from DB period last dose until Week 28. Median exposure to DB treatment was 24.50 weeks (minimum: 3.9 weeks; maximum: 160.4 weeks).
- DB Period: Placebo: Participants received placebo matched to macitentan dose levels during the DB treatment period. Participants who prematurely discontinued DB study treatment prior to Week 28 but did not withdraw consent were asked to enter PTOP from DB period last dose until Week 28. Median exposure to DB treatment was 44 weeks (minimum: 4 weeks; maximum: 147.9 weeks).
- Open Label (OL) Period: DB Macitentan: Participants who were treated with macitentan in the DB period and had reached the target dose of macitentan 75 mg and completed the DB period as per protocol were considered eligible to transition into the 104-week OL period and they continued macitentan 75 mg tablet orally QD from end of double blind treatment (EODBT) until study termination. Participants who experienced a clinical worsening event confirmed by the clinical event committee (CEC), were allowed to transition to the OL period at any time after Week 28. Median exposure to OL treatment was 72 weeks (minimum: 8.1 weeks; maximum: 84.6 weeks).
- OL Period: DB Placebo: Participants who were treated with placebo in the DB period and had completed the DB period as per protocol were considered eligible to transition into the 104-week OL period and were up-titrated to the target dose of macitentan 75 mg (macitentan 10 mg for 4 weeks, followed by macitentan 37.5 mg for another 4 weeks). Participants who experienced a clinical worsening event confirmed by the CEC, were allowed to transition to the OL period at any time after Week 28. Median exposure to OL treatment was 72 weeks (minimum: 8.1 weeks; maximum: 84.6 weeks).
Period: DB Period: Day 1 up to EODBT
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo | Open Label (OL) Period: DB Macitentan | OL Period: DB Placebo
Started | 64 | 63 | 0 | 0
Completed | 1 | 1 | 0 | 0
Not Completed | 63 | 62 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0
Not completed — Physician Decision | 8 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 4 | 0 | 0
Not completed — Study Terminated by Sponsor | 41 | 52 | 0 | 0
Not completed — Other | 8 | 5 | 0 | 0
Period: OL Period:Day 1 Upto End of OL Treatment
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo | Open Label (OL) Period: DB Macitentan | OL Period: DB Placebo
Started | 0 | 0 | 1 (Completed DB period) | 6 (1 participant who completed DB period + 5 participants who had CEC-confirmed clinical worsening event after DB period discontinuation)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 6
Not completed — Study Terminated by Sponsor | 0 | 0 | 1 | 5
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo | Total
Number analyzed (Participants) | 64 | 63 | 127
Age, Customized [Count of Participants; unit: Participants]
  Adults (18-64 years) | 23 | 33 | 56
  From 65 to 75 years | 32 | 26 | 58
  Over 75 years | 9 | 4 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 42 | 79
  Male | 27 | 21 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 59 | 58 | 117
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 18 | 26 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 42 | 34 | 76
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 4 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 0 | 1 | 1
  AUSTRALIA | 1 | 1 | 2
  BULGARIA | 1 | 2 | 3
  CHINA | 7 | 10 | 17
  CZECH REPUBLIC | 3 | 1 | 4
  DENMARK | 1 | 1 | 2
  FRANCE | 2 | 0 | 2
  GERMANY | 7 | 4 | 11
  HUNGARY | 1 | 1 | 2
  ISRAEL | 1 | 0 | 1
  ITALY | 3 | 1 | 4
  JAPAN | 5 | 9 | 14
  LITHUANIA | 0 | 1 | 1
  MEXICO | 2 | 2 | 4
  POLAND | 4 | 5 | 9
  PORTUGAL | 0 | 3 | 3
  ROMANIA | 3 | 0 | 3
  RUSSIAN FEDERATION | 5 | 0 | 5
  SAUDI ARABIA | 1 | 1 | 2
  SINGAPORE | 1 | 0 | 1
  SLOVAKIA | 1 | 0 | 1
  SOUTH KOREA | 3 | 5 | 8
  SPAIN | 1 | 1 | 2
  TAIWAN | 1 | 1 | 2
  THAILAND | 1 | 1 | 2
  TURKEY | 2 | 4 | 6
  UNITED KINGDOM | 2 | 0 | 2
  UNITED STATES | 5 | 8 | 13
AgeContinuous [Mean (Standard Deviation); unit: years] | 64.7 (11.69) | 60.3 (12.84) | 62.5 (12.41)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 6-minute Walk Distance (6MWD) at Week 28
Description: Change from baseline in 6MWD as measured by 6-minute walk test (6MWT) at Week 28 was reported. The purpose of the 6MWT was to quantify exercise tolerance and capacity. This standardized test measured the distance an individual was able to walk over a total of six minutes on a hard, flat surface with no obstacles. The goal was for the individual to walk as far as possible in 6 minutes.
Time Frame: Baseline (Day 1), Week 28
Population: Full analysis set (FAS) included all randomized participants assigned to a study intervention and were analyzed according to the intervention they had been assigned to via interactive web response system (IWRS). Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo
Number analyzed (Participants) | 47 | 48
Meters | 9.7 (5.81) | 25.8 (5.78)
Statistical Analysis 1: Comparison: Double Blind (DB) Period: Macitentan vs DB Period: Placebo; Test type: Superiority; p = 0.974, MMRM; Least square mean = -16.1, 95% CI 2-sided [-32.34 to 0.16], Standard Error of Mean 8.20 — Least square mean and SE of the mean was estimated by mixed model repeated measurements method

2. Secondary Outcome: Time to First Clinical Event Committee (CEC) Confirmed Clinical Worsening up to End-of Double-blind-treatment (EODBT) Period
Description: Time (months) to first CEC-confirmed clinical worsening up to EODBT were reported. Clinical worsening was defined as the occurrence of at least one of the following events: 1) All-cause death; 2) Heart and/or lung transplantation; 3) Unplanned pulmonary hypertension (PH)-related hospitalization; 4) PH-related deterioration from baseline identified by at least one of the following: a) Persistent increase in World Health Organization functional class (WHO FC) that could not be explained by another cause (for example, viral infection); b) Persistent deterioration by at least 15 percent (%) in exercise capacity; as measured by the 6MWD; c) New or worsened signs or symptoms of right heart failure; 5) Rescue pulmonary endarterectomy (PEA) and/or balloon pulmonary angioplasty (BPA) procedure due to worsening of PH.
Time Frame: From Baseline (Day 1) up to EODBT: median 24.5 weeks (min 3.9 weeks; max 160.4 weeks) for macitentan, median 44 weeks (min 4 weeks; max 147.9 weeks) for placebo
Population: FAS included all randomized participants assigned to a study intervention and were analyzed according to the intervention they had been assigned to via IWRS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo
Number analyzed (Participants) | 64 | 63
Months | NA [19.0 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with events. | NA [NA to NA] — Median, upper and lower limit of 95% CI were not estimable due to low number of participants with events.

3. Secondary Outcome: Number of Participants With Improvement in World Health Organization Functional Class (WHO FC) From Baseline to Week 28
Description: Number of participants with improvement in WHO FC from baseline to Week 28 were reported. Improvement (decrease) in WHO FC from baseline to Week 28 was calculated for each participant. WHO FC test was used to assess disease severity. Four functional classes (FC) were defined from FC I (no limitation of physical activity) to FC IV (inability to carry out any physical activity without symptoms). For the analysis purpose, these WHO FC class values were transformed to a scale with scores ranged from 1 to 4; where a score of 1 corresponded to WHO FC Class I and a score of 4 corresponded to WHO FC Class IV. The higher scores indicate greater symptom severity or worse impact. Improvement was considered when a participant changed from a higher class to a lower class.
Time Frame: From Baseline (Day 1) up to Week 28
Population: FAS included all randomized participants assigned to a study intervention and were analyzed according to the intervention they had been assigned to via IWRS. Here, 'N' (number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo
Number analyzed (Participants) | 37 | 43
Participants | 7 | 6

4. Secondary Outcome: Change From Baseline to Week 28 in Pulmonary Arterial Hypertension - Symptoms and Impact (PAH-SYMPACT) - Cardiopulmonary Symptom Domain Score
Description: The cardiopulmonary symptoms domain consisted of 6 items: shortness of breath, fatigue, lack of energy, swelling in ankles or legs, swelling in stomach area and cough and were reported on a 5-point Likert scale from 0 (no symptom at all) to 4 (very severe symptoms), with higher score indicating more symptom. The symptoms part of the PAH-SYMPACT was administered daily over a 7-day period. The recall period of symptom items was the last 24 hours. The mean individual symptom item score was determined for each of the 6 items and a domain score was calculated by summing the mean individual symptom item scores and dividing by the number of items, ranged from 0=no cardiopulmonary symptoms to 4=severe cardiopulmonary symptoms. A higher score indicated more severe symptoms experienced.
Time Frame: From Baseline (Day 1) up to Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo
Number analyzed (Participants) | 28 | 35
score on a scale | -0.089 (0.5856) | -0.060 (0.3767)

5. Secondary Outcome: Change From Baseline to Week 28 in PAH-SYMPACT - Cardiovascular Symptom Domain Score
Description: The cardiovascular symptoms domain consisted of 5 items: heart palpitations (fluttering), rapid heartbeat, chest pain, chest tightness, and lightheadedness and were reported on a 5-point Likert scale ranged from 0 (no symptoms at al) to 4 (very severe symptoms), with high score indicating more symptom. The symptoms part of PAH-SYMPACT was administered daily over a 7-day period. The recall period of symptom items was the last 24 hours. An average Cardiovascular Symptoms domain score was determined based on the daily scores of the 5 items. The mean individual symptom item score was determined for each of the 5 items and a domain score was calculated by summing the mean individual symptom item scores and dividing by the number of items, ranged from 0=no cardiovascular symptoms to 4=severe cardiovascular symptoms. Higher score indicated more severe symptoms experienced.
Time Frame: From Baseline (Day 1) up to Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo
Number analyzed (Participants) | 28 | 35
Score on a scale | -0.141 (0.4530) | -0.101 (0.2818)

6. Secondary Outcome: Change From Baseline to Week 28 in Euro Quality of Life-5-Dimension-5-Level (EQ-5D-5L) Utility Score and Visual Analog Scale (VAS) Score
Description: The EQ-5D-5L was a generic measure of health status. The EQ-5D-5L consisted of 2 parts: EQ-5D-5L utility score (descriptive system) and VAS score. EQ-5D-5L descriptive system consisted of 5-item questionnaire that assessed 5 domains including mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each questionnaire had 5 response levels: 1 =no problems, 2 =slight problems, 3 =moderate problems, 4 =severe problems and 5 =extreme problems. The scores for the 5 questionnaires were used to compute a single utility score which ranged from 0 to 1, where higher score indicated better health state and lower score indicated worse health state. EQ-5D-5L VAS rated current health state on a vertical scale with a score ranged from 0 (worst imaginable health state) to 100 (best imaginable health state), higher scores indicated a better health state.
Time Frame: From Baseline (Day 1) up to Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo
Number analyzed (Participants) | 29 | 33
Score on a scale
  Utility score | 0.0472 (0.26700) | 0.0050 (0.15010)
  VAS score | 5.0 (17.65) | 1.6 (11.97)

7. Secondary Outcome: Change From Baseline to Week 28 in Accelerometer-assessed Proportion of Time Spent in Moderate to Vigorous Physical Activity
Description: Change from baseline to Week 28 in accelerometer-assessed proportion of time spent in moderate to vigorous physical activity were assessed. Daily life physical activity of participant was assessed using accelerometer which was provided to the participant at screening and was worn daily during waking hours up to Week 28. For each scheduled visit, the 14 days prior to the visit were considered as the assessment period for physical activity. To be considered evaluable for a given timepoint, actigraphy variables should have been measured for at least 7 complete days (consecutive or not). A complete day is defined as a record of at least 7 waking hours of data. Proportion of time spent in moderate to vigorous physical activity was the estimated number of minutes spent in moderate or higher physical activity as calculated using the Staudenmayer '15 technique as proportion of the total minutes of algorithmically detected wear time and excluding the minutes that fall within a sleep period.
Time Frame: From Baseline (Day 1) up to Week 28
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percent of minutes per day
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo
Number analyzed (Participants) | 28 | 33
Percent of minutes per day | 0.821 (3.9249) | -0.833 (4.5160)

ADVERSE EVENTS:
Time Frame: DB period:DB Day 1 to 30 days post EODBT (median exposure[ME]:24.5 weeks[wks], [min 3.9 wks; max 160.4 wks] on macitentan, ME:44 wks [min 4 wks; max 147.9 wks] on placebo); OL period: OL Day 1 to study termination (ME:72 wks [min 8.1 wks; max 84.6 wks]).
Description: Safety analysis was based on safety analysis set which included all participants who received at least one dose of study intervention in this study and were analysed according to the intervention they actually received.
Groups:
- Open Label (OL) Period: DB Macitentan: Participants who were treated with macitentan in the DB period and had reached the target dose of macitentan 75 mg and completed the DB period as per protocol were considered eligible to transition into the 104-week OL period and they continued macitentan 75 mg tablet orally QD from EODBT until study termination. Participants who experienced a clinical worsening event confirmed by the CEC, were allowed to transition to the OL period at any time after Week 28. Median exposure to OL treatment was 72 weeks (minimum: 8.1 weeks; maximum: 84.6 weeks).
Arm/Group | Double Blind (DB) Period: Macitentan | DB Period: Placebo | Open Label (OL) Period: DB Macitentan | OL Period: DB Placebo
All-Cause Mortality (participants affected / at risk) | 1/64 | 0/63 | 0/1 | 0/6
Serious Adverse Events (participants affected / at risk) | 17/64 | 14/63 | 0/1 | 4/6
Other Adverse Events (participants affected / at risk) | 47/64 | 38/63 | 1/1 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB) Period: Macitentan (N=64) | DB Period: Placebo (N=63) | Open Label (OL) Period: DB Macitentan (N=1) | OL Period: DB Placebo (N=6)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Right Ventricular Failure (Cardiac disorders) | 1 | 0 | 0 | 1
Sinus Node Dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large Intestine Polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative Hypertension (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Fluid Retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Renal Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Transient Ischaemic Attack (Nervous system disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urge Incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Abnormal Uterine Bleeding (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 0 | 2
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Ovarian Cystectomy (Surgical and medical procedures) | 0 | 1 | 0 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0
Post Thrombotic Syndrome (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Double Blind (DB) Period: Macitentan (N=64) | DB Period: Placebo (N=63) | Open Label (OL) Period: DB Macitentan (N=1) | OL Period: DB Placebo (N=6)
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 0 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 6 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 4 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 3 | 0 | 0
Oedema Peripheral (General disorders) | 18 | 5 | 0 | 1
Pyrexia (General disorders) | 4 | 3 | 0 | 0
Swelling (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 4 | 0 | 0
Covid-19 (Infections and infestations) | 15 | 14 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 8 | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 4 | 0 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0
Haemoglobin Decreased (Investigations) | 7 | 0 | 0 | 1
Fluid Retention (Metabolism and nutrition disorders) | 4 | 0 | 0 | 0
Iron Deficiency (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0 | 1
Dizziness (Nervous system disorders) | 5 | 3 | 0 | 0
Headache (Nervous system disorders) | 9 | 10 | 0 | 1
Memory Impairment (Nervous system disorders) | 0 | 1 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 5 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 1 | 0 | 0
Hypotension (Vascular disorders) | 9 | 1 | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of participants analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04271475/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-18): https://cdn.clinicaltrials.gov/large-docs/75/NCT04271475/SAP_001.pdf